CLINICAL TRIAL: NCT03704571
Title: A Predictive Model for Inadequate Bowel Preparation: Development and Validation With a Randomized Controlled Trial
Brief Title: A Predictive Model for Inadequate Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018SDU-QILU-G111
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Bowel Preparation
Keywords: adenoma; bowel preparation; colonoscopy; predictive model; randomized controlled trial
MeSH Terms: conditions — Adenoma | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Group (Experimental): In the tailored group, high-risk patients are instructed to drink the first 2 L of Polyethylene Glycol (PEG) at 19:00-21:00 hours on the day before colonoscopy at a rate of 250 ml every 15 min. On the day of the procedure, they take another 2 L PEG 4-6 h before colonoscopy. The low-risk patients were given a standard dose of 2 L PEG 4-6 h before colonoscopy.
  Interventions: Drug: Polyethylene Glycol
- Control Group (Active Comparator): In the control group, all the patients drink single dose of 2 l Polyethylene Glycol (PEG) 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Interventions: Drug: Polyethylene Glycol

INTERVENTIONS:
Drug: Polyethylene Glycol — In the Tailored group, high-risk people are given intensified bowel preparation regimens, low-risk people are given routine regimens.
  In the control group, all the patients are given routine regimens.

SUMMARY:
We aimed to develop a predictive model of inadequate bowel preparation and to further validate it by a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years undergoing colonoscopy

Exclusion Criteria:

* known or suspected bowel obstruction, stricture or perforation
* compromised swallowing reflex or mental status
* severe chronic renal failure(creatinine clearance < 30 ml/min)
* severe congestive heart failure (New York Heart Association class III or IV)
* uncontrolled hypertension (systolic blood pressure > 170 mm Hg, diastolic blood pressure > 100 mm Hg)
* dehydration
* disturbance of electrolytes
* pregnancy or lactation
* hemodynamically unstable
* unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | 10 months
  The quality of bowel preparation is evaluated using BBPS.

SECONDARY OUTCOMES:
Adenoma Detection Rate | 10 months
  The proportion of patients from whom at least one adenoma can be detected.
Polyp Detection Rate | 10 months
  The proportion of patients from whom at least one polyp can be detected.
Adverse Events | 10 months
  Including nausea, bloating, stomachache, vomiting, vertigo and belching and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China